CLINICAL TRIAL: NCT06873347
Title: Electrical Fingerprint: Comparison of Characteristic Patterns of Different Surgical Interventions Based on Electrosurgical Unit Data
Brief Title: Electrosurgical Intervention Analysis: Comparing Procedure Patterns
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Erbe Elektromedizin GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MT_ERBE Data Logger
Record Dates: First submitted 2025-01-15; First posted 2025-03-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Procedure type: Procedures:
  * Supra cervical hysterectomy (+/- salpingectomy)
  * Total hysterectomy
  * Breast conserving surgeries: b-plastic + periareolar mastopexy (+/- Sentinel lymphonodectomy, SLNE)
  * Breast conserving surgeries: segmental resection (+/- SLNE)
  Data will be collected among patients who undergo surgery at the Department of Women's Health independently of this study.
  Interventions: Device: Procedure type
- Unknown

INTERVENTIONS:
Device: Procedure type — • Patients undergoing one of the following surgeries:
  * Supra cervical hysterectomy
  * Total hysterectomy
  * Breast conserving surgeries: B-plastic + periareolar mastopexy
  * Breast conserving surgeries: segmental resection
  Groups: Procedure type
Device:  — • A dataset from procedure types other than the above mentioned to the type "unknown" is assigned to this type.
  Groups: Unknown

SUMMARY:
The purpose of this prospective, single center study is to verify the hypothesis that each type of intervention creates a specific data pattern like a digital "fingerprint". This fingerprint offers the possibility to identify specific workflows of surgical procedures but also to differentiate between them, what can be used for training purposes. The following clinical study is not covered by the MDR regulation since we do not investigate performance or safety of a device but collect and assign electrical data only.

DETAILED DESCRIPTION:
The Erbe ESU VIO 3 provides electrical measurement data with high accuracy and time resolution. With the availability of the Erbe ECB Data Transmitter it is possible to record electrical data from the VIO 3 during clinical procedures, which open up a variety of possibilities for enhancing clinical workflows.

For this purpose, the VIO 3 will be connected via ECB (Erbe communication bus) interface with the "Data Transmitter". Using the software implemented by Erbe on the "Data transmitter", electrical data - generated during electrosurgical interventions - are recorded, forwarded via LAN, WLAN or LTE and stored in the Azure Cloud. These data do not contain any patient information and will be only used for the stated study objective.

In future, based on the analyses of electrosurgical device data users could benefit from e.g. continuous training as well as self enhancement/reflection by electrosurgical information offered during or after a surgical procedure. A first step to reach this goal is to build up a database containing electrosurgical data of different surgical interventions, to identify the electrosurgical "fingerprint" of each intervention and to detect different patterns between them. Therefore, the purpose of this study is to record electrosurgical data and to verify the hypothesis that each type of intervention creates a specific data pattern like a digital "fingerprint".

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent
* Patients undergoing one of the following surgeries:

  * Supra cervical hysterectomy
  * Total hysterectomy
  * Breast conserving surgeries: B-plastic + periareolar mastopexy
  * Breast conserving surgeries: segmental resection

Exclusion Criteria:

* Expected lack of patient compliance or inability of the patient to understand the purpose of the clinical trial
* Lack of patient consent
* Surgery under local anaesthesia
* Robot-Assisted Surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted as a single-center study with patient recruitment among patients who visit the Department of Women's Health. No patients must be recruited only for the purpose of this study. Data will be collected among patients who undergo surgery at the Department of Women's Health independently of this study. The prospective, single center study is designed as a pilot study. A case number estimate is not possible. The aim is to include a total of about 160 patients in the pilot study.
  Procedure Number of cases Supra cervical hysterectomy 40 Total hysterectomy 40 B-plastic + periareolar mastopexy 40 Segmental resection 40
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Identification of Unique Electrosurgical Data Patterns ("Digital Fingerprints") for Surgical Procedures | During surgery and post-procedure analysis (data collection over 12 months)
  The study aims to determine whether different types of surgical interventions generate distinct electrosurgical data patterns. The accuracy of assigning recorded electrosurgical data to the correct surgical procedure type will be evaluated.
  Data Source: Electrosurgical signals recorded by the Erbe ECB Data Transmitter and VIO 3 system, stored in the Erbe Cloud for analysis.
  Measurement Method:
  * Each dataset will be classified into one of the predefined procedure types or as "unknown."
  * The classification algorithm must achieve at least 80% accuracy in correctly identifying procedure types.
  * The classification algorithm must achieve at least 80% accuracy in assigning procedures outside the predefined types to the "unknown" category.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Krämer, Prof. Dr., Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany